CLINICAL TRIAL: NCT04934904
Title: The Treatment of Acute Gastrointestinal Injury Via Ultrasound-guided Erector Spinae Plane Block - a Prospective, Single-center, Randomized, Controlled Trial
Brief Title: The Treatment of Acute Gastrointestinal Injury Via Ultrasound-guided Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-KY-032-03
Record Dates: First submitted 2021-06-03; First posted 2021-06-22 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2021-10

CONDITIONS: Gastrointestinal Disease
Keywords: Acute gastrointestinal injury; Erector spinal muscle plane block; Ropivacaine
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Experimental Group:
  On the basis of the clinical routine treatment of AGI in severe patients (gastrointestinal dynamic drugs, traditional Chinese drugs and physical rehabilitation therapy), the ultrasound-guided erector spinae plane block intervention is given.
  Controlled Group:
  Normal Treatment.
Masking Description: This study adopted a randomized, open, blank control design, and did not blind researchers, patients or clinicians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): On the basis of the clinical routine treatment of AGI in severe patients, the Experimental Group will receives ultrasound-guided erector spinae plane block with routine treatment of AGI for 7 days or until transferring to the general ward.
  Interventions: Drug: Ropivacaine injection
- Controlled Group (No Intervention): the routine clinical treatment of AGI is given to severe patients, such as gastrointestinal dynamic drugs, traditional Chinese drugs and physical rehabilitation therapy

INTERVENTIONS:
Drug: Ropivacaine injection — On the first day of inclusion, performed T8 bilateral ultrasound-guided erector spinae plane block and indwelling tube will be left + 0.375% ropivacaine 20ml to both sides. Patients will be given injections every 12 h for 7 days.
  Other Names: ropivacaine
  Arms: Experimental Group

SUMMARY:
In this single-center, randomized, parallel control clinical trial, patients will be randomly assigned to two groups. The treatment group receives ultrasound-guided erector spinae plane block with routine treatment of Acute Gastrointestinal Injury (AGI) for 7 days or until transferred to the general ward, while the control group only receives routine treatment of AGI. The primary outcome is the cure and remission rate of AGI.

DETAILED DESCRIPTION:
Detailed Description:

Study title: The treatment of Acute Gastrointestinal Injury via ultrasound-guided erector spinae plane block - a prospective, single-center, randomized, controlled trial

Principal Investigator: Professor Wang Hua, Department of Critical Care Unit, Zhujiang Hospital of Southern Medical University

Study subjects: Patients age from 18 to 80 with AGI Ⅱ or greater

Study phase: Investigator Initiated Trial(IIT)

Primary objectives:

To evaluate whether ultrasound-guided erector spinae plane block can reduce the grade of AGI , and improve the cure and remission rate of AGI.

Experimental Group:

On the basis of routine clinical treatment, the ultrasound-guided erector spinae plane block intervention is given. On the first day enrolled, patients are performed with ultrasound-guided erector spinae plane block and cannula will be placed on T8 bilaterally. 0.375% ropivacaine of 20ml is injected separately to both sides with 2ml per hour. Injection is performed twice a day for 7 days or until transferred to the general ward.

Controlled Group:

The patients will receive the clinical routine treatment according of AGI recommended by the 2012 European Society of Critical Care Medicine guidelines, with a uniform nutritional strategy(gastrointestinal dynamic drugs, traditional Chinese drugs and physical rehabilitation therapy).

Course: 7 days Sample size: 100 Sites: 1

Primary endpoints:

1. the cure rate of AGI
2. the remission rate of AGI

Secondary endpoints:

1. critical ill scores
2. Gastrointestinal function indicators
3. The inflammatory indicators
4. the lactic acid(Lac)
5. cross-sectional area of pyloric antrum(AS) with ultrasound
6. width of the colons with abdominal X ray or CT
7. the 28-day mortality
8. gastrointestinal dysfunction and duration (GIF)

Additional endpoints:

1. The length of stay in ICU
2. The total days of hospitalization

ELIGIBILITY:
Inclusion Criteria:

1. AGI are diagnosed according to the diagnostic criteria proposed by European Society Intensive Care Medicine (ESICM) in 2012 and the AGI grade great than or equal to II.
2. Age 18-80 years.
3. Expected length of stay longer than 3 days.

Exclusion Criteria:

1. Mean arterial pressure is still less than 65 millimeter of Mercury (mmHg) treated with rehydration and vasoactive agents, or with the dosage of norepinephrine more than 0.5ug/kg/min.
2. Heart rates are less than 50 beats per minute or moderate and severe atrioventricular block without pacemaker.
3. Primary gastrointestinal disease such as mechanical intestinal obstruction, massive hemorrhage of gastrointestinal tract and gastrointestinal perforation.
4. Severe trauma of chest, abdomen or back. gastrointestinal tract surgery history.
5. Neuromuscular disorders.
6. Drug addiction, alcohol abuse, opioid or amphetamine dependence, or mental disorders.
7. Pregnancy.
8. Brain dead.
9. Malignant tumor, or end-stage cachexia.
10. With contraindications of the erector spinae plane block (ESPB), such as local infection, Spinal diseases or immobilization.
11. Allergy to local anesthetics.
12. Significant abnormalities in blood coagulation parameters.
13. Without written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
the cure rate of AGI | on the day3
  the cure rate of AGI on the day3
the cure rate of AGI | on the day7
  the cure rate of AGI on the day7
the remission rate of AGI | on the day3
  the remission rate of AGI on the day3
the remission rate of AGI | on the day7
  the remission rate of AGI on the day7

SECONDARY OUTCOMES:
Acute Physiology and Chronic Health Evaluation(APACHE II) | on the day 0,1,3 and 7
  measuring endpoints include:
  body temperature
  mean arterial pressure (MAP)
  heart rate (HR)
  respiratory rate (RR)
  fraction of inspiration O2 (FIO2)
  potential of hydrogen (PH)
  Na+
  K+
  serum creatinine (SCr)
  hematocrit (Hct%)
  white blood cell (WBC)
  Age
  immunosuppression before/after surgery or serious organ dysfunction
  (Higher score means a worse outcome.)
Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score | on the day 0,1,3 and 7
  SOFA score evaluate status of the following organ systems separately:
  (Higher score means a worse outcome.)
  1. Respiration Partial Pressure of Oxygen/Fraction of Inspiration O2 (PaO2/FiO2)
  2. Coagulation Platelets
  3. Liver Bilirubin
  4. Circulatory Mean arterial pressure
  5. Central Nervous System Glasgow coma score
  6. Renal Creatinine (or urine output)
the intraperitoneal pressure(IAP) | on the day 0,1,3 and 7
  Gastrointestinal function indicators
abdominal perfusion pressure(AAP) | on the day 0,1,3 and 7
  Gastrointestinal function indicators
total gastric residual volume(GRVs) | on the day 0,1,3 and 7
  Gastrointestinal function indicators
feeding dose | on the day 0,1,3 and 7
  Gastrointestinal function indicators
Gastrointestinal dysfunction and duration(GIF) | on the day 0,1,3 and 7
  1. fasting(score 1 point)
  2. reflux(score 2 points)
  3. gastrointestinal decompression(1 point)
  4. Gastric retention(2 points)
  5. abdominal distension(2 points)
  6. abdominal pain(2 points)
  7. diarrhea(2 points)
  8. hypoactive bowel sounds(1 point)
  9. bowel sounds disappear(2 points)
  10. constipation(2 points)
  The mentioned indicators will be combined to report GIF in score.
  Grade 0 (Normal) : 0 score
  Grade 1 (Mild) : 1~4 score
  Grade 2 (Medium) : 5~9 score
  Grade 3 (Serious) : >10 score
Width of the colons | on the day 0,1,3 and 7
  width of the right colons with abdominal X ray or CT
White Blood Cell(WBC) | on the day 0,1,3 and 7
  The inflammatory indicators
Interleukin-6(IL-6) | on the day 0,1,3 and 7
  The inflammatory indicators
Cross-sectional area of pyloric antrum(AS) | on the day 0,1,3 and 7
  cross-sectional area of pyloric antrum(AS) with ultrasound
Lymphocyte (LYM) | on the day 0,1,3 and 7
  The inflammatory indicators
Neutral Granular Cell(NEUT) | on the day 0,1,3 and 7
  The inflammatory indicators
Procalcitonin (PCT) | on the day 0,1,3 and 7
  The inflammatory indicators
Hypersensitive C Reactive Protein(HSCRP) | on the day 0,1,3 and 7
  The inflammatory indicators
The lactic acid(Lac) | on the day 0,1,3 and 7
  the serum level of the lactic
The 28-day mortality | From enrolled to 28 days or the termination date
  the 28-day mortality
The length of stay in ICU | on the day 28 or through study completion
  From the date of ICU admission to transfered out.
The total days of hospitalization | on the day 28 or through study completion
  from hospital admission to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Wang, MD,PhD, Principal Investigator — Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No